CLINICAL TRIAL: NCT04445974
Title: Can a Brief Body-functionality Writing Intervention Improve Body Image in Individuals Living With a Skin Condition? A Randomised Control Trial
Brief Title: Testing a Body-functionality Intervention for Body Image in Individuals With Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 165478
Record Dates: First submitted 2020-06-16; First posted 2020-06-24 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Body Image; Psychological Distress; Dermatologic Disease; Quality of Life
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Intervention Model Description: This study is an online single-blinded Randonmised Control Trial, which contains acceptability and feasibility components.
Who Masked: Participant
Masking Description: Participants will not be told whether they have been allocated to intervention or control condition until the end of the study. The control condition is a series of creative writing tasks, which are framed as an intervention within the introduction to the first task. This replicates previous RCTs of the same intervention in different populations (Alleva et al., 2015).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expand Your Horizons: More than my skin (Active Comparator): Participants allocated to the intervention condition will be asked to follow the adapted instructions for 'Expand Your Horizon'. Participants will be asked to complete three 15 min writing exercises over approximately six days. Participants who complete the first exercise on Qualtrics will be sent links to and asked to complete the second and third writing exercises.
  Interventions: Behavioral: Expand your horizons: More than my skin
- Control writing activity (Experimental): Participants in the control condition will be asked to complete three 15 minute creative writing exercises online via Qualtucs over approximately six days. Participants completing the first writing exercise will be sent links to the second and third writing exercises.
  Interventions: Behavioral: Creative writing activities

INTERVENTIONS:
Behavioral: Expand your horizons: More than my skin — 'Expand Your Horizon' is a self-help intervention which uses writing exercises to help individuals with poor body image practice focusing on their body-functionality rather than their physical appearance (Alleva et al., 2015). The materials for 'Expand Your Horizon' are freely available (Alleva et al., 2015), and permission has been granted to use and adapt the materials in this research. 'Expand Your Horizon' comprises of three 15 min writing exercises, typically completed over approximately six days. The intervention materials have been adapted for use with a population with skin diseases, and modified to use gender neutral language. Adaptions were made in consultation with experts by experience. The changes were reviewed and approved by the first author of the original intervention to ensure the materials were in keeping with the original intervention.
  Arms: Expand Your Horizons: More than my skin
Behavioral: Creative writing activities — In line with previous studies examining 'Expand Your Horizon' the active control condition will involve creative writing tasks (Alleva et al., 2015). Participants in the intervention condition will complete three 15 minute creative writing exercises, completed over six days.
  Arms: Control writing activity

SUMMARY:
'Expand Your Horizons', a self-help writing intervention that seeks to train individuals to focus on what their body can do (functionality) rather than what it looks like (appearance), has produced promising results in improving body image. However, it has not been adapted and trialled in populations with conditions affecting skin appearance. This research therefore seeks to evaluate the potential for 'Expand Your Horizons' to (1) improve body image, as measured by body and functionality appreciation; and (2) improve skin-specific outcome, as measure by skin-shame, dermatology and quality of life, in a population with dermatological conditions, using a Randomised Control Trail.

DETAILED DESCRIPTION:
Method of sampling/recruitment:

Recruitment from community sample, including: The University staff and student volunteers lists; Psychology undergraduate credit systems, Social media/forums; Charities; Research recruitment platforms, and a mailing lists.

Sample size:

An apriori power analysis, based on an ANCOVA, with a medium effect for the primary outcome (body appreciation) indicated a sample of 128 would be needed to achieve 80% power. Assuming an attrition rate of 50%, the total number of participants required will be 256.

In line with recommendations for evaluating interventions, we will include an internal pilot whereby we review the recruitment progress (completion) about 3 months into the trial and could then consider whether we need to make any minor or major adjustments to the recruitment strategy or study. If these substantial changes are needed, the pilot component will be written up and analysed separately to inform the next phase.

Procedure:

Time-point 1: Participants asked to read information sheet and provide consent. Participants will then be asked to complete the demographic measures and provide information on their skin condition(s). Participants will then complete baseline measures of trait body appreciation, body functionality, and, skin-specific quality of life, appearance anxiety with the order of these questionnaires counterbalanced. The online system will then randomly allocate individual meeting the exclusion criteria to either 'Expand Your Horizon' or an active control, at a ratio of 1:1. Participants will then be asked to complete the first writing activity and complete state measures

Time-point 2 (approximately 2 days later): Participants asked to complete the second writing exercise, and rate their state measures.

Time-point 3 (approximately 1 week later): Participants will be asked to complete the final writing task, before completing state measures and repeating the outcome measures given at baseline. Participants in both conditions will then be asked to provide feedback on the intervention.

Time-point 4 (One month later): Participants will be asked to repeat the outcome measures. Participants will then be shown the debrief screen and told which group they were in. Participants in the control condition will be offered a link to the intervention.

Analytic strategy:

The data will be initially assessed to check whether they meet the assumptions of the statistical tests used.

Descriptive statistics will then be used to describe the sample, and to summarise information on attrition at each point of the study and feedback on the intervention. Demographic and skin disease-history variables will be assessed for covariance using t-tests, ANOVAs and bivariate correlations as appropriate.

To assess whether randomisation of allocation to groups (intervention vs control) has been effective, t-tests and ANOVAs will be used, as appropriate, to compare demographics baseline measures.

T-tests will also be used to compare the levels of skin-specific appearance satisfaction, appearance satisfaction and body-functionality satisfaction between participants in both the intervention and control condition. This will include both intention-to-treat and completer analyses.

The effectiveness of the intervention will be tested using a series of between group ANCOVAs.

The number of participants showing reliable and clinical change on measures of anxiety and skin-specific quality of life will also be calculated for each group.

Change over time (Pre, post, one month follow up) for each group will be assessed using a repeated measures ANOVA. If any significant covariates, are identified ANCOVAs will be used instead.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with dermatological condition (including conditions that affect the skin, hair and/or nails). This includes, but is not limited to, acne, eczema, alopecia, psoriasis, vitiligo, rosacea, dermatitis, hyperpigmentation, hidradenitis suppurativa (HS), hyperhidrosis, hirsutism, neurofibromatosis, onychomycosis, melasma, cysts, herpes, ichthyosis, and lichen sclerosus.
* Individuals self-reporting that their body image is affected by their skin condition.
* Sufficient English to complete the measures and writing exercises
* Access to the internet.

Exclusion Criteria:

* As the focus of this research is on skin disease, individuals living with visible differences as a consequence of trauma (e.g. scarring from burns or scarring from traumatic injury) are not eligible to participate in this study.
* Individuals who do not feel their body image is affected by having a dermatological condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Change in body appreciation | Baseline to 1 week
  The Body Appreciation Scale 2 (BAS-2, Tylka & Wood-Barcalow, 2015) will be used to measure body appreciation and contains 10 items, and will be used to measure trait levels of body appreciation. Each item is rated on a scale of 1 (never) to 5 (always). The average score is calculated by adding each item and divided by 10, and can range between 1 and 5 with higher numbers indicating higher levels of body appreciation.
Change in body functionality appreciation | Baseline to 1 week
  The Functionality Appreciation Scale (FAS: Alleva, Tylka, & Van Diest, 2017) will be used to measure body functionality appreciation. The FAS comprises of seven questions, and will be used to assess participants' trait levels of appreciation for their bodies' functionality (Appendix L). Each item is rated on a scale from 1 (strongly disagree) to 5 (strongly agree). The average score is calculated by adding each item and dividing by 7, and can range between 1 and 5 with higher numbers indicating higher levels of function appreciation.

SECONDARY OUTCOMES:
Change in dermatology specific quality of life | Baseline to 1 week
  The Dermatology Quality of Life Index (DLQI: Finlay & Khan, 1994) will be used to measure the impact of skin-conditions on participants' quality of life (Appendix M). The DLQI contains 10 questions scored from 0 (not at all/not relevant) to 3 (very much). Total scores range from 0 to 30, with lower scores indicating greater skin-specific quality of life.
Change in dermatology specific quality of life at follow up | Baseline to 1 month
  The Dermatology Quality of Life Index (DLQI: Finlay & Khan, 1994) will be used to measure the impact of skin-conditions on participants' quality of life (Appendix M). The DLQI contains 10 questions scored from 0 (not at all/not relevant) to 3 (very much). Total scores range from 0 to 30, with lower scores indicating greater skin-specific quality of life.
Chance in skin-specific shame | Baseline to 1 week
  The Skin Shame Scale (SSS: Scott, 2004) will be used to measure levels of skin-specific shame. The SSS contains 24 items, which are rated on a scale from 1 (never) to 5 (always). Total scores can range from 24 to 120, with higher score indicating greater levels of shame.
Chance in skin-specific shame at follow up | Baseline to 1 month
  The Skin Shame Scale (SSS: Scott, 2004) will be used to measure levels of skin-specific shame. The SSS contains 24 items, which are rated on a scale from 1 (never) to 5 (always). Total scores can range from 24 to 120, with higher score indicating greater levels of shame.
Change in appearance anxiety | Baseline to 1 week
  The Appearance Anxiety Index (AAI: Veale et al., 2014) will be used to measure appearance anxiety. The AAI contains 10 questions focused on cognitive and behavioural components of appearance-related anxiety, including avoidance and threat monitoring. Each item is scored on a five point Likert scale from 0 (not at all) to 4 (all the time). Total scores can range from 0 to 40, with higher scores indicating a greater level of appearance-related anxiety.
Change in appearance anxiety at follow up | Baseline to 1 month
  The Appearance Anxiety Index (AAI: Veale et al., 2014) will be used to measure appearance anxiety. The AAI contains 10 questions focused on cognitive and behavioural components of appearance-related anxiety, including avoidance and threat monitoring. Each item is scored on a five point Likert scale from 0 (not at all) to 4 (all the time). Total scores can range from 0 to 40, with higher scores indicating a greater level of appearance-related anxiety.
State appearance satisfaction | Day 1
  After writing exercise 1, participants will also be asked to rate their state satisfaction with their appearance on a 100 point visual analogue scale (100 = extremely satisfied and 0 = extremely dissatisfied).
State appearance satisfaction | Day 3 (approximately)
  After writing exercise 2, participants will also be asked to rate their state satisfaction with their appearance on a 100 point visual analogue scale (100 = extremely satisfied and 0 = extremely dissatisfied).
State appearance satisfaction | 1 week
  After writing exercise 3, participants will also be asked to rate their state satisfaction with their appearance on a 100 point visual analogue scale (100 = extremely satisfied and 0 = extremely dissatisfied).
State skin appearance satisfaction | Day 1
  After writing task 1, participants will also be asked to rate their satisfaction with their state skin appearance on a 100 point visual analogue scale (100 = extremely satisfied and 0 = extremely dissatisfied).
State skin appearance satisfaction | Day 3 (approximately)
  After writing task 2, participants will also be asked to rate their satisfaction with their state skin appearance on a 100 point visual analogue scale (100 = extremely satisfied and 0 = extremely dissatisfied).
State skin appearance satisfaction | 1 week
  After writing task 3, participants will also be asked to rate their satisfaction with their state skin appearance on a 100 point visual analogue scale (100 = extremely satisfied and 0 = extremely dissatisfied).
State functionality satisfaction | Day 1
  After writing task 1, participants will also be asked to rate their state satisfaction with their body functionality on a 100 point visual analogue scale (100 = extremely satisfied and 0 = extremely dissatisfied).
State functionality satisfaction | Day 3 (approximately)
  After writing task 2, participants will also be asked to rate their state satisfaction with their body functionality on a 100 point visual analogue scale (100 = extremely satisfied and 0 = extremely dissatisfied).
State functionality satisfaction | 1 week
  After writing task 3, participants will also be asked to rate their state satisfaction with their body functionality on a 100 point visual analogue scale (100 = extremely satisfied and 0 = extremely dissatisfied).
Change in body appreciation at follow up | Baseline to 1 month
  The Body Appreciation Scale 2 (BAS-2, Tylka & Wood-Barcalow, 2015) will be used to measure body appreciation and contains 10 items, and will be used to measure trait levels of body appreciation. Each item is rated on a scale of 1 (never) to 5 (always). The average score is calculated by adding each item and divided by 10, and can range between 1 and 5 with higher numbers indicating higher levels of body appreciation.
Change in body functionality appreciation at follow up | Baseline to 1 month
  The Functionality Appreciation Scale (FAS: Alleva, Tylka, & Van Diest, 2017) will be used to measure body functionality appreciation. The FAS comprises of seven questions, and will be used to assess participants' trait levels of appreciation for their bodies' functionality (Appendix L). Each item is rated on a scale from 1 (strongly disagree) to 5 (strongly agree). The average score is calculated by adding each item and dividing by 7, and can range between 1 and 5 with higher numbers indicating higher levels of function appreciation.

OTHER OUTCOMES:
Intervention evaluation | 1 week
  Participants in the functionality intervention will be asked to complete a series of questions about their experience of the intervention, and given the option to add any further comments in a free text box.
Adherence | Through study completion (on average 1 week)
  Adherence will be assessed by reviewing the content of participants writing and time-spent on the exercises and word count. Participant entries will also be rated, on a three-point scale, whether the content of participants writing conforms to the given instructions; if there is no relevant content, it will be scored 0, if instructions are partially followed, it will score 1, and if instruction are fully followed it will score a 2.
  to identify inappropriate responses. Previous studies evaluating the intervention have reported minimal information about how adherence was assessed.
Attrition | Through study completion (on average 1 week)
  The number of participants that drop out across the study

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Overton, PhD, Principal Investigator — University of Sheffield
Locations (1):
- Department of Psychology, University of Sheffield, Sheffield, Choose Province, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participants will be asked as part of the consent form whether they would be willing for their anonymised data to be available to other researchers. Data won't be shared for participants who do not consent to this. Sharing of the remaining data will depend on sufficient participants consenting to this to not compromise anonymity or outcomes.

REFERENCES:
- [Background] Alleva JM, Martijn C, Van Breukelen GJ, Jansen A, Karos K. Expand Your Horizon: A programme that improves body image and reduces self-objectification by training women to focus on body functionality. Body Image. 2015 Sep;15:81-9. doi: 10.1016/j.bodyim.2015.07.001. Epub 2015 Aug 14. PMID 26280376
- [Background] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Background] Alleva JM, Tylka TL, Kroon Van Diest AM. The Functionality Appreciation Scale (FAS): Development and psychometric evaluation in U.S. community women and men. Body Image. 2017 Dec;23:28-44. doi: 10.1016/j.bodyim.2017.07.008. Epub 2017 Aug 17. PMID 28822275
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Scott, C. (2004). Understanding psychodermatological distress: constructing a skin shame scale (Doctoral dissertation, University of Sheffield, UK). Retrieved from http://etheses.whiterose.ac.uk/14863/1/412462.pdf
- [Background] Veale D, Eshkevari E, Kanakam N, Ellison N, Costa A, Werner T. The Appearance Anxiety Inventory: validation of a process measure in the treatment of body dysmorphic disorder. Behav Cogn Psychother. 2014 Sep;42(5):605-16. doi: 10.1017/S1352465813000556. Epub 2013 Jul 3. PMID 23823485
- [Derived] Adkins KV, Overton PG, Thompson AR. A brief online writing intervention improves positive body image in adults living with dermatological conditions. Front Med (Lausanne). 2022 Dec 21;9:1064012. doi: 10.3389/fmed.2022.1064012. eCollection 2022. PMID 36619619